CLINICAL TRIAL: NCT02136056
Title: Effects of a Self-management Course for Adults on Sick-leave; Outcomes in Registry Based Measures of Return to Work and Questionnaire Based Measures of Well-being and Quality of Life
Brief Title: Effects of a Self-management Course for Adults on Sick-leave
Acronym: jos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); VIVE - The Danish Center for Social Science Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: auh_JOS_sfi-01
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2017-12-08 (Actual); Status verified 2016-09

CONDITIONS: Workers on Sick-leave, Insured by The Danish Welfare State
Keywords: Sick-leave; Return to work; Self-management; Self-efficacy; Quality of Life and Well-being; Motivation
MeSH Terms: interventions — Self-Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Self-management program (SMP) (Experimental): Participants in the experimental group receive six weekly group-sessions of self-management and patient education; specifically targeting self-management of the return to work process and disease symptoms.
  Interventions: Behavioral: Self-management program (SMP)
- Treatment as usual (No Intervention): Participants in the control-group receive standard rehabilitation care and follow-up in the job-center.

INTERVENTIONS:
Behavioral: Self-management program (SMP) — A self-management course
  Other Names: Stanford patient education
  Arms: Self-management program (SMP)

SUMMARY:
The purpose of the current study is to determine the efficacy of a self-management course for workers on sick-leave as an add-on to standard rehabilitation care and follow-up (treatment as usual). Outcomes are registry based measures of return to work, and questionnaire based measures of well-being and quality of life.

We thus, hypothesize that the program will improve workers return to work rates and self-reported/psychological well-being.

DETAILED DESCRIPTION:
The intervention course is a Danish adaptation of The Chronic Disease Self-Management Program (CDSMP), tailored towards workers on sick-leave. The original program has been developed by The Stanford Patient Education Research Center. The translation and adaptation has been conducted by The Danish Committee for Health Education.

Previous studies have examined the program with respect to specific chronic diseases (e.g., Arthritis), quality of life, well-being and health-care utilization, though non-otherwise specified workers on sick-leave and return work have not been examined before.

The framework of CDSMP is social-cognitive learning theory in which self-efficacy plays a central role.

ELIGIBILITY:
Inclusion Criteria:

* Insured persons who receive sick-leave compensation from the Danish State
* Persons who are listed as sick from a job
* Persons who have been categorized as "2 - risk" or "3 - chronic" case by the job-center
* The health problem reflects a chronic or a long-term condition
* The person acknowledges a chronic or long-term condition
* The person wants to work with his or her condition
* The person wants to return to work
* The person volunteers to participate

Exclusion Criteria:

* Persons who are listed sick for more than 16 weeks
* Persons who are categorized as "1 - easy" by the job-center
* The person does not understand or speak danish
* History or signs of aggressive behavior and violence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Return to work, duration | Weekly from baseline till 1 year follow-up
  DREAM-registry (supported by the Danish Ministry of Employment) combined with income/employment information from e-income (supported by the Danish Tax Authorities).
Well-being and Quality of life | up to 5 month follow-up
  WHO-5 Well-being and WHO Quality of Life/Satisfaction items (Bech, 2012)

SECONDARY OUTCOMES:
Common mental disorders | Baseline, post-intervention and 4,5 month follow-up
  The CMDQ questionnaire i based on SCL-90 (Symptom Checklist) and measures somatization, health-anxiety, depression, anxiety and alcohol consumption (Christensen et al., 2005)
Disease self-efficacy scale | Baseline, post-intervention and 4,5 month follow-up
  The University of Washington Self-efficacy scale, 6 item version (Amtmann et al., 2012)
Self-regulation (return to work) | Baseline, post-intervention and 4,5 month follow-up
  Return to work self-regulation questionnaire, measuring internalization of reasons for trying to return to work; adapted from the Treatment Self-regulation Questionnaire (Levesque et al., 2007)
Self-management scale | Baseline, post-intervention and 4,5 month follow-up
  A measure of six cognitive strategies which are taught at the course (Lorig et al., 1996)
Illness Perception questionnaire | Baseline, post-intervention and 4,5 month follow-up
  A measure of 8 items measuring the threat of illness or disease (B-IPQ; Broadbent, Petrie, Main & Weinman, 2006)

OTHER OUTCOMES:
Health-care utilization | Baseline, post-intervention and 4,5 month follow-up
  Items that measure utilization of health-care consultation (Lorig et al., 1996)
Medicine consumption | Baseline, post-intervention and 4,5 month follow-up
  Generic items that measure consumption of medicines such as anti-depressants and anxiety medicine, use of pain killers and sleep pills
Adherence to treatment | Baseline, post-intervention and 4,5 month follow-up
  Adherence to disease specific treatment (inspired by the MMAS-4; Morisky & DiMatteo, 2011)
Common symptoms | Baseline, post-intervention and 4.5 month follow-up
  Pain, breath, being tired, sleep quality; measured by VAS scales (Lorig et al., 1996)
Decisional Balance (return to work) | Baseline, post-intervention and 4,5 month follow-up
  Generic items that measures how the advantages and disadvantages of returning to work are balanced (Franche & Krause, 2002)
Return to work expectations | Baseline, post-intervention and 4,5 month follow-up
  Generic items that measure expectations about returning to work (Niewenhuiksen, Noordik, van Dijk & van der Klink. 2013; Schultz et al., 20014)

CONTACTS AND LOCATIONS:
Overall Officials: Martin H Olesen, PhD, Study Director — Aarhus University and Aarhus University Hospital; Jan Høgelund, PhD, Study Chair — VIVE - The Danish Center for Social Science Research; Mimi Y Mehlsen, PhD, Principal Investigator — University of Aarhus
Locations (1):
- The Danish Comitee for Health Education, Copenhagen, Denmark

REFERENCES:
- [Background] Bech, P. Clinical Psychometrics. Oxford: Wiley-Blackwell, 2012.
- [Background] Christensen KS, Fink P, Toft T, Frostholm L, Ornbol E, Olesen F. A brief case-finding questionnaire for common mental disorders: the CMDQ. Fam Pract. 2005 Aug;22(4):448-57. doi: 10.1093/fampra/cmi025. Epub 2005 Apr 6. PMID 15814580
- [Background] Bjorner JB, Damsgaard MT, Watt T, Groenvold M. Tests of data quality, scaling assumptions, and reliability of the Danish SF-36. J Clin Epidemiol. 1998 Nov;51(11):1001-11. doi: 10.1016/s0895-4356(98)00092-4. PMID 9817118
- [Background] Amtmann D, Bamer AM, Cook KF, Askew RL, Noonan VK, Brockway JA. University of Washington self-efficacy scale: a new self-efficacy scale for people with disabilities. Arch Phys Med Rehabil. 2012 Oct;93(10):1757-65. doi: 10.1016/j.apmr.2012.05.001. Epub 2012 May 7. PMID 22575393
- [Background] Franche RL, Krause N. Readiness for return to work following injury or illness: conceptualizing the interpersonal impact of health care, workplace, and insurance factors. J Occup Rehabil. 2002 Dec;12(4):233-56. doi: 10.1023/a:1020270407044. PMID 12389476
- [Background] Nieuwenhuijsen K, Noordik E, van Dijk FJ, van der Klink JJ. Return to work perceptions and actual return to work in workers with common mental disorders. J Occup Rehabil. 2013 Jun;23(2):290-9. doi: 10.1007/s10926-012-9389-6. PMID 23124685
- [Background] Schultz IZ, Crook J, Meloche GR, Berkowitz J, Milner R, Zuberbier OA, Meloche W. Psychosocial factors predictive of occupational low back disability: towards development of a return-to-work model. Pain. 2004 Jan;107(1-2):77-85. doi: 10.1016/j.pain.2003.09.019. PMID 14715392
- [Background] Levesque CS, Williams GC, Elliot D, Pickering MA, Bodenhamer B, Finley PJ. Validating the theoretical structure of the Treatment Self-Regulation Questionnaire (TSRQ) across three different health behaviors. Health Educ Res. 2007 Oct;22(5):691-702. doi: 10.1093/her/cyl148. Epub 2006 Nov 30. PMID 17138613
- [Background] Lorig, K., Stwart, A., Ritter, P., Gonzales, V., Laurent, D., & Lynch, J. Outcome measures for health education and other health care interventions. Thousand Oaks, CA: Sage Publications. 1996.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Marks R, Allegrante JP, Lorig K. A review and synthesis of research evidence for self-efficacy-enhancing interventions for reducing chronic disability: implications for health education practice (part I). Health Promot Pract. 2005 Jan;6(1):37-43. doi: 10.1177/1524839904266790. PMID 15574526
- [Background] Marks R, Allegrante JP, Lorig K. A review and synthesis of research evidence for self-efficacy-enhancing interventions for reducing chronic disability: implications for health education practice (part II). Health Promot Pract. 2005 Apr;6(2):148-56. doi: 10.1177/1524839904266792. PMID 15855284
- [Background] Lorig K, Laurent DD, Plant K, Krishnan E, Ritter PL. The components of action planning and their associations with behavior and health outcomes. Chronic Illn. 2014 Mar;10(1):50-9. doi: 10.1177/1742395313495572. Epub 2013 Jul 9. PMID 23838837
- [Background] Broadbent E, Petrie KJ, Main J, Weinman J. The brief illness perception questionnaire. J Psychosom Res. 2006 Jun;60(6):631-7. doi: 10.1016/j.jpsychores.2005.10.020. PMID 16731240
- [Background] Morisky DE, DiMatteo MR. Improving the measurement of self-reported medication nonadherence: response to authors. J Clin Epidemiol. 2011 Mar;64(3):255-7; discussion 258-63. doi: 10.1016/j.jclinepi.2010.09.002. Epub 2010 Dec 8. No abstract available. PMID 21144706
- See also: Web-page that describes the course — http://www.patientuddannelse.info/jos.aspx